CLINICAL TRIAL: NCT04675463
Title: An Open Label, Single-center, Prospective, Interventional Pilot Study to Evaluate the Effects of Inhaled Budesonide-formoterol-glycopyrronium and Formoterol-glycopyrronium in Moderate-to-severe Chronic Obstructive Pulmonary Disease
Brief Title: The Effects of Inhaled Budesonide-formoterol-glycopyrronium in Moderate-to-severe COPD
Acronym: OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ShiYue Li (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCT-19-20271
Record Dates: First submitted 2020-11-27; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide/Glycopyrronium/Formoterol arm (Other): 52 weeks treatment
  Interventions: Drug: BGF Inhalation Aerosphere
- Glycopyrronium/Formoterol arm (Other): 52 weeks treatment
  Interventions: Drug: GFF Inhalation Aerosphere

INTERVENTIONS:
Drug: BGF Inhalation Aerosphere — Budesonide/Glycopyrronium/Formoterol: 160/7.2/4.8/ puff, twice daily with two puffs per time
  Other Names: Breztri
  Arms: Budesonide/Glycopyrronium/Formoterol arm
Drug: GFF Inhalation Aerosphere — Glycopyrronium/Formoterol: 7.2/4.8 per puff, twice daily with two puffs per time
  Other Names: Bevespi
  Arms: Glycopyrronium/Formoterol arm

SUMMARY:
The fixed-dose combination product Budesonide/Glycopyrronium/Formoterol Fumarate Inhalation Aerosol, BGF pMDI and dual combination product Glycopyrronium/Formoterol Fumarate Inhalation Aerosol , GFF pMDI are developed for maintenance treatment for patients with COPD.

There are still some unmet medical needs and evidence gaps in COPD therapy, such as could BGF Inhalation Aerosphere reverse the disease progression such like airway-remodelling? Could BGF Inhalation Aerosphere reduce inflammation in small airways? Before differences proven between medication groups, pilot study is needed.

This 52 weeks, Single-center, prospective, interventional pilot study could help discovering intervention effect of BGF and GFF on small airways through OCT measurement, which would show outcome of AEROSPHERE™ Delivery Technology on COPD patients.

DETAILED DESCRIPTION:
The subjects eligible for this study will receive a 52-week of BGF or GFF treatment, and a 30 days follow-up telephone call after the last study drug dose.

ELIGIBILITY:
Inclusion Criteria:

* With capability of communicating via oral conversation or written documents and signing informed consent.
* With capability of receiving and participating in study related auxiliary examinations.
* Age: 40-80 yrs, both male and female, with or without smoking history, receiving treatment in community hospitals or outpatient department in general hospitals
* GOLD Stage II-III COPD: FEV1/FVC<70% and FEV1 45-80% predicted (about 1/3 subjects in 45%-50%), measured 20min after 400μg salbutamol inhalation
* With stable COPD (no COPD exacerbation during the latest 4 weeks prior to the recruitment) and irregular use of inhalation therapy, or regular use of inhalation therapy but no more than 2 weeks. Subject is willing and, in the opinion of the investigator, able to adjust current COPD therapy, as required by the protocol.

Exclusion Criteria:

* Subjects are participating in other clinical research or have completed another clinical research within 3 months prior to screening.
* Significant diseases or conditions other than COPD. A significant disease or condition is defined as a disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the patients' ability to participate in the study
* Patients with clinical diagnosis of lung cancer, bronchiectasis, pneumoconiosis, or other single restricted ventilation.
* Severe cardiovascular, neural, hepatic, renal and hematologic diseases or malignancies that may interfere with the operation of the study.
* Patients with prostatic hyperplasia or bladder neck obstruction with significant symptoms, or narrow angle glaucoma
* Patients have a current and history diagnosis of asthma, or who have a blood eosinophil count ≥600/mm3 (0.6×109/L).
* Patients with active pulmonary tuberculosis
* Patients with life-threatening pulmonary embolism, α1-antitrypsin deficiency, or cystic fibrosis
* History of pneumonectomy.
* COPD exacerbation in 4 weeks prior to the first visit (V1), or hospitalization and/or antibiotic application and/or oral or intravenous glucocorticosteroids application is required during screening stage.
* Long-term oxygen therapy, frequent use of glucocorticosteroids orally or intravenously (prednisone>10mg/d), or long-term use of antibiotics.
* Women who are pregnant or lactating or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
* Planned hospitalization or blood donation during the trial.
* Known hypersensitivity or intolerance to trial drugs.
* History of chronic alcohol or drug abuse, or any other conditions that may impact compliance.
* With contraindications to undergo bronchoscopy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The effect of BGF and GFF on inner luminal area change | 12 months
  Change from baseline in the inner luminal area of the 7th to 9th generation bronchi (Ai7-9) at month 12 measured by Endobronchial optical coherence tomography (EB-OCT)

SECONDARY OUTCOMES:
The effect of BGF and GFF on luminal diameter change | 12 months
  •Change from baseline in mean luminal diameter of the 7th to 9th generation bronchi (Dmean7-9) at month 12 measured by EB-OCT
The effect of BGF and GFF on airway wall area change | 12 months
  •Change from baseline in airway wall area percentage of the 7th to 9th generation bronchi (Aw%7-9) at month 12 measured by EB-OCT
The effect of BGF and GFF on resonant frequency | 12 months
  •Change from baseline in resonant frequency (Fres) at month 6 and 12 measured by impulse oscillometry (IOS)
The effect of BGF and GFF on peripheral airway resistance | 12 months
  •Change from baseline in peripheral airway resistance (R5-R20) at month 6 and 12 measured by IOS
The effect of BGF and GFF on lung function including FEV1, FVC,FEV1% | 12 months
  •Change from baseline in trough FEV1, FVC and FEV1% at month 6 and 12 measured by spirometry

OTHER OUTCOMES:
Exploratory Objective: change of Quality of life | 12 months
  • the effects of BGF and GFF in improving quality of life measured by St. George's Respiratory Questionnaire (SGRQ),Scores range from 0 to 100, with higher scores indicating more limitations.
Exploratory Objective: change of emphysema | 12 months
  •the effects of BGF and GFF in reducing emphysema measured by Computer Tomography(CT)
Exploratory Objective: TNF-α | 12 months
  • the effects of BGF and GFF in ameliorating COPD inflammation measured by TNF-α in sputum
Exploratory Objective: IL-1β | 12 months
  • the effects of BGF and GFF in ameliorating COPD inflammation measured by IL-1β in sputum
Exploratory Objective: MMP-8 | 12 months
  • the effects of BGF and GFF in ameliorating COPD inflammation measured by MMP-8 in sputum
Exploratory Objective: MMP-12 | 12 months
  • the effects of BGF and GFF in ameliorating COPD inflammation measured by MMP-12 in sputum

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Doctor, Principal Investigator — Guangzhou Institute of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Diseases, Guangzhou, Guangdong, China